CLINICAL TRIAL: NCT05172128
Title: Effect of Blueberry Supplementation on Alzheimer's Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00108907
Record Dates: First submitted 2021-12-09; First posted 2021-12-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: MCI; biomarkers; memory loss
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blueberry supplementation (Experimental): All participants will receive 18 grams lyophilized blueberry supplement mixed with water twice daily for 12 weeks.
  Interventions: Dietary Supplement: lyophilized blueberry supplement

INTERVENTIONS:
Dietary Supplement: lyophilized blueberry supplement — lyophilized blueberry supplement bid

SUMMARY:
The purpose of this study is to study the effects of blueberries on neuronal, glial, and pathology blood biomarkers in Mild Cognitive Impairment (MCI) and to estimate sample size for future confirmatory studies. The blood biomarkers to be measured are Neurofilament light (NfL), glial fibrillary acidic protein (GFAP), Aß40, Aß42, p-tau181, and cytokines, using an ultra-sensitive state-of-the-art immunoassay.

DETAILED DESCRIPTION:
After determining subject eligibility and after subjects have abstained from consuming all berry fruits (including red wine) for 2 weeks, subjects will have blood drawn for biomarkers and will then will undergo 12 weeks of blueberry supplementation in the form of 18 grams lyophilized blueberry powder mixed with water and taken twice daily with meals. All subjects will be asked to abstain from berry fruits (including red wine) for the duration of the 12 week trial. Subjects will receive telephone calls at 4 and 8 weeks to check compliance as well as concomitant medications and adverse events and then all subjects will return at 12 weeks for a repeat biomarker blood draw. Plasma NfL, GFAP, Aβ40, Aβ42, p-tau181, and cytokine biomarker assays will be done using the Quanterix SR-X instrument, a new, state-of-the-art digital immunoassay platform employing Simoa technology, which enables the detection and quantification of biomarkers previously difficult or impossible to measure.

ELIGIBILITY:
Inclusion Criteria:

1. 55 to 85 years old inclusive
2. Meets criteria for amnestic Mild Cognitive Impairment defined by education adjusted performance on the Wechsler Memory Scale (WMS) III Logical Memory delayed recall score and clinical evaluation.
3. Medically stable

Exclusion Criteria:

1. Dementia
2. Significant confounding active neurological/psychiatric disease
3. Participation in an experimental investigational drug trial in the past 30 days
4. Unwilling to restrict consumption of anthocyanin-rich foods
5. Inability to complete cognitive testing (e.g. significant visual or hearing impairment)
6. Allergy or intolerance to blueberries
7. Significant gastrointestinal disorders or surgery that influences digestion and absorption
8. Presence of unstable, acutely symptomatic, or life-limiting illness
9. Women of childbearing potential

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murali Doraiswamy, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller MG, Hamilton DA, Joseph JA, Shukitt-Hale B. Dietary blueberry improves cognition among older adults in a randomized, double-blind, placebo-controlled trial. Eur J Nutr. 2018 Apr;57(3):1169-1180. doi: 10.1007/s00394-017-1400-8. Epub 2017 Mar 10. PMID 28283823
- [Background] Wang S, Cui Y, Wang C, Xie W, Ma L, Zhu J, Zhang Y, Dang R, Wang D, Wu Y, Wu Q. Protective Effects of Dietary Supplementation with a Combination of Nutrients in a Transgenic Mouse Model of Alzheimer's Disease. PLoS One. 2015 Nov 25;10(11):e0143135. doi: 10.1371/journal.pone.0143135. eCollection 2015. PMID 26606074
- [Background] Jeong HR, Jo YN, Jeong JH, Kim HJ, Kim MJ, Heo HJ. Blueberry (Vaccinium virgatum) leaf extracts protect against Abeta-induced cytotoxicity and cognitive impairment. J Med Food. 2013 Nov;16(11):968-76. doi: 10.1089/jmf.2013.2881. Epub 2013 Oct 11. PMID 24117094
- [Background] Brewer GJ, Torricelli JR, Lindsey AL, Kunz EZ, Neuman A, Fisher DR, Joseph JA. Age-related toxicity of amyloid-beta associated with increased pERK and pCREB in primary hippocampal neurons: reversal by blueberry extract. J Nutr Biochem. 2010 Oct;21(10):991-8. doi: 10.1016/j.jnutbio.2009.08.005. Epub 2009 Dec 1. PMID 19954954
- [Background] Ou Y, Hu H, Wang Z, Xu W, Tan L, et al. Plasma neurofilament light as a longitudinal biomarker of neurodegeneration in Alzheimer's disease. Brain Science Advances. 2019;5(2):94-105.

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Blueberry Supplementation: single arm blueberry supplementation
Period: Overall Study
Arm/Group | Single Arm Blueberry Supplementation
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Blueberry Supplementation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.20 (5.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Education [Mean (Standard Deviation); unit: years] | 18.10 (2.15)
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE (Mini Mental State Examination) is a 30 question test measuring several cognitive domains including memory, orientation, attention and language. The test is scored on a scale of 0 to 30 with higher scores indicating better cognitive function. MCI range for study inclusion was 23 or higher.
  units on a scale | 27.20 (2.15)
Weschler Logical Memory Delay [Mean (Standard Deviation); unit: units on a scale] — The Weschler Logical memory test involves reading a story to the subject and asking them to recall the story verbatim immediately after presentation as well as after a 20-30 minute delay. The story has 25 discrete details and recall score ranges from 0-25. The lower the score, the greater the cognitive impairment. MCI is defined by a delayed Logical memory score of <12 (if ≥16 years education) or ≤9 (if 8-15 years education).
  units on a scale | 4.80 (3.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Neurofilament Light (NfL) Levels as Measured by Blood Biomarker Assay
Description: Change in NfL level from baseline to 12 weeks as measured by blood biomarker assay in pg/mL
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 10
pg/mL
  Baseline | 30.09 (4.64)
  12 weeks | 44.25 (16.85)
Statistical Analysis 1: Comparison: Blueberry Supplementation; Test type: Other; p > 0.05, t-test, 2 sided; Paired t-test comparing baseline value to endpoint value revealed a p-value of 0.80

2. Primary Outcome: Change in Blood Glial Fibrillary Acidic Protein (GFAP) Levels as Measured by Blood Biomarker Assay
Description: Change in blood glial fibrillary acidic protein (GFAP) levels from baseline to 12 weeks as measured by blood biomarker assay in pg/mL
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 10
pg/mL
  Baseline | 239.86 (31.15)
  12 weeks | 234.27 (26.98)
Statistical Analysis 1: Comparison: Blueberry Supplementation; Test type: Other; p > 0.05, t-test, 2 sided

3. Primary Outcome: Change in Blood Amyloid Beta 42/40 as Measured by Blood Biomarker Assay
Description: Change in blood Amyloid beta 42/40 ratio (Aβ42 divided by Aβ40) from baseline to 12 weeks as measured by blood biomarker assay. Lower ratios increase likelihood of AD pathology.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 10
ratio
  Baseline | .050 (.002)
  12 weeks | .050 (.002)
Statistical Analysis 1: Comparison: Blueberry Supplementation; Test type: Other; p > 0.05, t-test, 2 sided

4. Primary Outcome: Change in P-tau 181 as Measured by Blood Biomarker Assay
Description: Change in p-tau 181 from baseline to 12 weeks as measured by blood biomarker assay in pg/mL
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 10
pg/mL
  Baseline | 37.24 (3.31)
  12 weeks | 38.04 (2.58)
Statistical Analysis 1: Comparison: Blueberry Supplementation; Test type: Other; p > 0.05, t-test, 2 sided

5. Primary Outcome: Change in Blood Interleukin-6 (IL-6) Levels as Measured by Blood Biomarker Assay
Time Frame: Baseline, 12 weeks
Population: Data not collected.
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 0

6. Primary Outcome: Change in Tumor Necrosis Factor (TNF-alpha) Levels as Measured by Blood Biomarker Assay
Time Frame: Baseline, 12 weeks
Population: Data not collected.
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 0

7. Primary Outcome: Change in Brain-derived Neurotrophic Factor (BDNF)
Description: Change in brain-derived neurotrophic factor (BDNF) from baseline to 12 weeks in pg/mL
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Blueberry Supplementation
Number analyzed (Participants) | 10
pg/mL
  Baseline | 1685.48 (480.43)
  12 weeks | 1850.15 (436.63)
Statistical Analysis 1: Comparison: Blueberry Supplementation; Test type: Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Blueberry Supplementation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blueberry Supplementation (N=10)
altered mental status (Nervous system disorders) | 1 (1) — Subject admitted to hospital overnight for altered mental status and generalized weakness. Workup negative for stroke but TIA could not be ruled out. Symptoms resolved by discharge.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blueberry Supplementation (N=10)
constipation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1) — 1 episode
tremor/weakness (Nervous system disorders) | 1 (1) — transient
Covid infection (Infections and infestations) | 1 (1)
hematemesis (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT05172128/Prot_SAP_000.pdf